CLINICAL TRIAL: NCT02657746
Title: Control of Blood Pressure and Risk Attenuation-Bangladesh, Pakistan and Sri Lanka (COBRA-BPS)
Brief Title: Primary Care Strategies to Reduce High Blood Pressure: A Cluster Randomized Trial in Rural Bangladesh, Pakistan and Sri Lanka
Acronym: COBRA-BPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Aga Khan University (Other); University of Kelaniya (Other)
Responsible Party: Principal Investigator, Professor Tazeen Jafar, Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MR/N006178/1
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Hypertension
Keywords: blood pressure monitoring; high blood pressure; cardiovascular disease; Antihypertensive agents; Non-pharmacological treatment; community health care workers; cost-effectiveness
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- usual care (No Intervention): Usual care comprises existing services for hypertension control in the community without any additional training
- multi-component interventions (Experimental): : The multi-component interventions (MCI) is comprised of all the following five components: 1) home health education (HHE) by government community health workers (CHWs), plus 2) blood pressure (BP) monitoring and stepped-up referral to a trained general practitioner (GP) using a checklist, plus 3) training public and private providers in management of hypertension and using a checklist, plus 4) designating hypertension triage counter and hypertension care coordinators in government clinics, plus 5) a financing model to compensate for additional health services and provide subsides to low income individuals with poorly controlled hypertension.
  Interventions: Other: multi-component interventions

INTERVENTIONS:
Other: multi-component interventions — The multi-component interventions (MCI) is comprised of all the following five components: 1) home health education (HHE) by government community health workers (CHWs), plus 2) blood pressure (BP) monitoring and stepped-up referral to a trained general practitioner (GP) using a checklist, plus 3) training public and private providers in management of hypertension and using a checklist, plus 4) designating hypertension triage counter and hypertension care coordinators in government clinics, plus 5) a financing model to compensate for additional health services and provide subsides to low income individuals with poorly controlled hypertension.
  Arms: multi-component interventions

SUMMARY:
Background: High blood pressure (BP) is the leading attributable risk for cardiovascular disease (CVD). In rural South Asia, hypertension remains to be a significant public health issue with sub-optimal rates of case finding and management. The goal of the full-scale study is to evaluate the effectiveness and cost-effectiveness of multicomponent primary care strategies on lowering blood pressure among adults with hypertension in rural communities in Bangladesh, Pakistan, and Sri Lanka.

Methods/Design: The mixed-methods, stratified cluster randomized controlled trial

Intervention: The multi-component interventions (MCI) is comprised of all the following five components: 1) home health education (HHE) by government community health workers (CHWs), plus 2) blood pressure (BP) monitoring and stepped-up referral to a trained general practitioner (GP) using a checklist, plus 3) training public and private providers in management of hypertension and using a checklist, plus 4) designating hypertension triage counter and hypertension care coordinators in government clinics, plus 5) a financing model to compensate for additional health services and provide subsides to low income individuals with poorly controlled hypertension.

Usual care: Will comprise existing services in the community without any additional training.

Participants: The trial will be conducted on 2550 individuals aged 40 years or older with hypertension (systolic BP ≥ 140 mm Hg or diastolic BP≥ 90 mm Hg, or on antihypertensive therapy) in 30 rural communities of Bangladesh, Pakistan and Sri Lanka. Out of the 2550 individuals, 420 with poorly controlled BP (Systolic BP≥160 mmHg or Diastolic BP≥100 mmHg) will be selected, 14 from each community, to investigate the effect of MCI on results from ambulatory BP monitoring.

Qualitative component: Stakeholders including policymakers, district managers, and community health workers, GPs, hypertensive individuals and family members in the identified clusters will be surveyed.

Outcome: The primary outcome will be change in systolic BP from baseline to follow-up at 24 months post randomization. The cost effectiveness outcome is the incremental cost of MCI per unit reduction in BP over the two year time period and in terms of incremental cost per CVD DALYs averted.

ELIGIBILITY:
Main study:

Inclusion Criteria:

1. Age≥ 40 years
2. Residing in the selected clusters
3. Hypertension defined either as:

   1. Persistently elevated BP (systolic BP ≥140 mm Hg or diastolic BP ≥90 mm Hg) from each set of last 2 of 3 readings from 2 separate days
   2. maintained on anti-hypertensive medications
4. Informed consent

Exclusion Criteria:

1. Permanently bed-ridden individuals too ill to commute to the clinic
2. Pregnancy, or individuals with advanced medical disease (on dialysis, liver failure, other systemic diseases)
3. Individuals that are mentally compromised and unable to give informed consent

Sub-study:

1) fulfill all criteria of main study and, 2) Persistently elevated systolic BP >160 mm Hg or diastolic BP >100 mm Hg from each set of 2 readings from 2 separate days

-

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2550 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Blood pressure reading:change in systolic blood pressure (SBP) from baseline to follow-up at 24 months post randomization. | Blood pressure (BP) will measured at baseline and then at 6-month intervals until 24 months after randomization

SECONDARY OUTCOMES:
Blood pressure reading:Blood Pressure(BP) controlled to target (Systolic BP <140 mm Hg and Diastolic BP <90 mm | at 6-month intervals over 24 months
Questionnaire:Composite outcome of death (all cause), or hospital admission due to coronary heart disease (CHD), heart failure, or stroke | 24 months
Questionnaire and EQ-5D-5L:Incremental cost per quality-adjusted life-year (QALY) gained from baseline to end of follow-up | 24 months
Morisky Medication Adherence Scale(MMAS):Change in antihypertensive medication adherence (Morisky score) | 24 months
Height and weight measurements:change in body mass index ( BMI) | 24 months
questionnaire:change dietary salt intake (urinary excretion) | 24 months
Questionnaire:change in prevalence of current smokers | 24 months
Questionnaire:incident diabetes | 24 months
Lipid panel: change in serum lipid levels | 24 months
questionnaire: change in INTERHEART cardiovascular disease (CVD) risk score | 24 months
Questionnaire:incidence of adverse outcomes (medication side effects, sick days absenteeism, low QALY between randomized groups). | 24 months
Questionnaire and serum creatinine:Change in estimated glomerular filtration rate (eGFR) | 24 months
Urine albumin:Change in urine albumin | 24 months
24 hours mean diastolic BP | 24 months
  Secondary outcome for the sub-study of 420 patients with poorly controlled BP at baseline
Daytime SBP/DBP | 24 months
  secondary outcome for the sub-study of 420 patients with poorly controlled BP at baseline
Night time SBP/DBP | 24 months
  Secondary outcome for the sub-study of 420 patients with poorly controlled BP at baseline
Dipping Pattern | 24 months
  Secondary outcome for the sub-study of 420 patients with poorly controlled BP at baseline
24 hour BP variability | 24 months
  Secondary outcome for the sub-study of 420 patients with poorly controlled BP at baseline
Questionnaire and EQ-5D-5L:Incremental cost per mm Hg BP reduction from baseline to end of follow-up at two years post randomization and incremental cost per projected cardiovascular disease ( CVD) disability adjusted life year (DALY) averted | information on healthcare cost will be collected at baseline and 24 months
incremental cost per mm Hg BP reduction from baseline to end of follow-up at 2 years post-randomization and incremental cost per projected CVD disability-adjusted life year (DALY) averted | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Tazeen H Jafar, MD,MPH, Principal Investigator — Duke-NUS Graduate Medical School

REFERENCES:
- [Derived] Feng L, Jehan I, de Silva HA, Naheed A, Khan AH, Kasturiratne A, Clemens JD, Lim CW, Hughes AD, Chaturvedi N, Jafar TH. Effect of a Multicomponent Intervention on Antihypertensive Medication Intensification in Rural South Asia: Post Hoc Analysis of a Cluster RCT. Am J Hypertens. 2021 Sep 22;34(9):981-988. doi: 10.1093/ajh/hpab072. PMID 34013966
- [Derived] Jafar TH, Gandhi M, de Silva HA, Jehan I, Naheed A, Finkelstein EA, Turner EL, Morisky D, Kasturiratne A, Khan AH, Clemens JD, Ebrahim S, Assam PN, Feng L; COBRA-BPS Study Group. A Community-Based Intervention for Managing Hypertension in Rural South Asia. N Engl J Med. 2020 Feb 20;382(8):717-726. doi: 10.1056/NEJMoa1911965. PMID 32074419
- [Derived] Perera M, de Silva CK, Tavajoh S, Kasturiratne A, Luke NV, Ediriweera DS, Ranasinha CD, Legido-Quigley H, de Silva HA, Jafar TH. Patient perspectives on hypertension management in health system of Sri Lanka: a qualitative study. BMJ Open. 2019 Oct 7;9(10):e031773. doi: 10.1136/bmjopen-2019-031773. PMID 31594895
- [Derived] Gandhi M, Assam PN, Turner EL, Morisky DE, Chan E, Jafar TH; COBRA-BPS Study Group. Statistical analysis plan for the control of blood pressure and risk attenuation-rural Bangladesh, Pakistan, Sri Lanka (COBRA-BPS) trial: a cluster randomized trial for a multicomponent intervention versus usual care in hypertensive patients. Trials. 2018 Nov 29;19(1):658. doi: 10.1186/s13063-018-3022-8. PMID 30486858
- [Derived] Feng L, de Silva HA, Jehan I, Naheed A, Kasturiratne A, Himani G, Hasnat MA, Jafar TH. Regional variation in chronic kidney disease and associated factors in hypertensive individuals in rural South Asia: findings from control of blood pressure and risk attenuation-Bangladesh, Pakistan and Sri Lanka. Nephrol Dial Transplant. 2019 Oct 1;34(10):1723-1730. doi: 10.1093/ndt/gfy184. PMID 29982770
- [Derived] Jafar TH, Gandhi M, Jehan I, Naheed A, de Silva HA, Shahab H, Alam D, Luke N, Wee Lim C; COBRA-BPS Study Group. Determinants of Uncontrolled Hypertension in Rural Communities in South Asia-Bangladesh, Pakistan, and Sri Lanka. Am J Hypertens. 2018 Oct 15;31(11):1205-1214. doi: 10.1093/ajh/hpy071. PMID 29701801
- [Derived] Jafar TH, Jehan I, de Silva HA, Naheed A, Gandhi M, Assam P, Finkelstein EA, Quigley HL, Bilger M, Khan AH, Clemens JD, Ebrahim S, Turner EL; for COBRA-BPS Study Group; Kasturiratne A. Multicomponent intervention versus usual care for management of hypertension in rural Bangladesh, Pakistan and Sri Lanka: study protocol for a cluster randomized controlled trial. Trials. 2017 Jun 12;18(1):272. doi: 10.1186/s13063-017-2018-0. PMID 28606184